CLINICAL TRIAL: NCT06183541
Title: Effects of Pericapsular Nerve Group (PENG) Block Applied for Analgesia on the Postoperative Process in Patients Undergoing Hip Fracture Surgery.
Brief Title: Effects of Pericapsular Nerve Group Block Applied in Patients Undergoing Hip Fracture Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeliha Alicikus, Assistant professor, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UERH-AR-ZT-03
Record Dates: First submitted 2023-12-03; First posted 2023-12-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hip Fractures; Pain, Postoperative
Keywords: PENG block; Anesthesia
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: This prospective randomised controlled study included a total of 70 patients aged 30-85 years who underwent hip fracture surgery under spinal anaesthesia. Patients were divided into two groups as PENG block and non-PENG block (control group).
Who Masked: Participant
Masking Description: Patients who underwent PENG block and those who did not undergo PENG block are randomly divided into two groups using the sealed envelope method. They are grouped as Group I: Those who received PENG block (n: 35) and Group II: Those who did not receive PENG block (control group) (n: 35).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG Block group (Active Comparator): PENG block group; USG probe is placed on the transverse plane medial to the anterior inferior iliac spine (AIIS), the medial end of the probe is placed on the superior pubic It is rotated approximately 45° counterclockwise to align it with the ramus. For the PENG block, an 80 mm block needle is placed in the fascial plane between the psoas tendon and pubic ramus and 20 ml of 0.5% bupivacaine is administered after spinal anesthesia,
  Interventions: Procedure: Pericapsular Nerve Group (PENG) Block
- Control group (Other): Control group; 10 ml 0.5% bupivacaine + 10 ml 2% lidocaine is infiltrated into the surgical area by the surgical team at the end of surgery
  Interventions: Procedure: Pericapsular Nerve Group (PENG) Block

INTERVENTIONS:
Procedure: Pericapsular Nerve Group (PENG) Block — Pericapsular nerve group (PENG) block The femoral nerve and obturator nerve terminal branches, which provide sensory innervation of the hip joint, are blocked, thus providing analgesia without creating a motor block.

SUMMARY:
In this study, it was aimed to compare the multimodal analgesia application or the pericapsular nerve group (PENG) block methods in patients undergoing hip surgery. The effectiveness and benefit rate of the PENG block in postoperative pain will be evaluated.

Postoperative pain, need for additional analgesia, range of motion of the hip joint, mobilization time, length of hospital time and adverse events in patients undergoing hip fracture surgery with and without PENG block will be investigated.

DETAILED DESCRIPTION:
This prospective randomised controlled study included a total of 70 patients aged 30-85 years who underwent hip fracture surgery under spinal anaesthesia. Patients were randomly divided into two groups using the sealed envelope method, Group I: those who received PENG block (n:35) and Group II:Those who did not receive PENG block (control group) (n: 35).

All patients will undergo hip fracture surgery by the same surgical team. Each patient will be informed about the procedure to be performed during anesthesia and surgery, and signed informed consent will be obtained before the procedure.Patients in Group I who will undergo the PENG block method; Before surgery, after spinal anesthesia, PENG block is performed under sterile conditions under ultrasonography guidance. With the patient supine, a 2-5 MHz, low-frequency, curvilinear probe is placed in the transverse plane medial to the anterior inferior iliac spine (AIIS), with the medial end of the probe rotated approximately 45° counterclockwise to align with the superior pubic ramus.

With the PENG block, an 80 mm block needle is placed in the fascial plane between the psoas tendon and the pubic ramus and 20 ml of 0.5% bupivacaine is administered.

As for the patients in Group II (control group); It is a routine practice at the end of surgery; 10 ml 0.5% bupivacaine + 10 ml 2% lidocaine is infiltrated into the surgical area by the surgical team.

For routine postoperative multimodal analgesia, intravenous PCA (patient controlled analgesia) was administered to patients in both groups with tramadol 50 mg at a basal rate of 10 mg / hour after loading (20 mg bolus dose + 30 minutes lock time) and paracetamol 10 mg / kg iv. (Given every 8 hours)

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo hip fracture surgery Women and men aged 30-85

Exclusion Criteria:

* Patients under 30 years old, over 85 years old
* American Society of Anesthesiology (ASA) IV,
* Those with cognitive impairment (alzheimer, dementia, delirium, etc.)
* Those with application site infection
* Those who are allergic to local anesthetic substances
* Patients are non-consenting patients.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score | 30 min, 12th, 24th and 48th hours in the postoperative period
  VAS pain score
Total opioid consumption | postoperative 48 hours
  Tramadol (mg)
mobilisation time | postoperative 24-48 hours
  take 5 steps with walker

SECONDARY OUTCOMES:
PENG block adverse events | between the time surgery starts and the 48th hour
  motor block, nerve damage, hypotension, bradycardia
length of hospital stay | between the time of hospitalization for the operation and discharge (day)
  day

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Tuncel, MD, Study Director — Umraniye Education and Research Hospita
Locations (2):
- Turkey (Türkiye) (2):
  - Umraniye Education and Research Hospital, Istanbul, Umraniye
  - UmraniyeERH, Istanbul, Umraniye

IPD SHARING:
Plan to Share IPD: No